CLINICAL TRIAL: NCT01962207
Title: A PHASE IIIB, OPEN, MULTI-CENTER STUDY TO EVALUATE THE LONG-TERM ANTIBODY PERSISTENCE AT 6, 7, 8, 9 AND 10 YEARS AFTER THE ADMINISTRATION OF ONE DOSE OF THE MENINGOCOCCAL CONJUGATE VACCINE MENACWY-TT VERSUS ONE DOSE OF MENINGITEC(REGISTERED) VACCINE OR ONE DOSE OF THE MENINGOCOCCAL POLYSACCHARIDE VACCINE MENCEVAX(REGISTERED) ACWY, AND TO EVALUATE THE SAFETY AND IMMUNOGENICITY OF A BOOSTER DOSE OF MENACWY-TT VACCINE ADMINISTERED 10 YEARS AFTER PRIMARY VACCINATION OF 1-10 YEAR OLD SUBJECTS WITH MENACWY-TT, MENINGITEC(REGISTERED) OR MENCEVAX(REGISTERED) ACWY.
Brief Title: The Long-term Antibody Persistence of MenACWY-TT Vaccine (PF-06866681) Versus Meningitec(Registered) or Mencevax(Registered) ACWY in Healthy Adolescents and Adults and a Booster Dose of MenACWY-TT Administered 10 Years Post Primary Vaccination
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MENACWY-TT-100; 2013-001549-15 (EudraCT Number); C0921004 (Other: Alias Study Number); 200171 (Other: Alias Study Number)
Record Dates: First submitted 2013-09-26; First posted 2013-10-14 (Estimated); Results first posted 2019-06-07 (Actual); Last update posted 2019-06-07 (Actual); Status verified 2019-03

CONDITIONS: Infections, Meningococcal
Keywords: 10 years Meningitec; Safety; booster response; Adolescents; Adults; Immunogenicity; Mencevax ACWY
MeSH Terms: conditions — Meningococcal Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ACWY<2 Group (Experimental): Subjects will receive a dose of MenACWY-TT 10 years after primary vaccination with MenACWY-TT.
  Interventions: Biological: Meningococcal vaccine GSK134612
- ACWY≥2 Group (Experimental): Subjects will receive a dose of MenACWY-TT 10 years after primary vaccination with MenACWY-TT.
  Interventions: Biological: Meningococcal vaccine GSK134612
- MenCCRM Group (Experimental): Subjects will receive a dose of MenACWY-TT 10 years after primary vaccination with Meningitec.
  Interventions: Biological: Meningococcal vaccine GSK134612
- MenPS Group (Experimental): Subjects will receive a dose of MenACWY-TT 10 years after primary vaccination with Mencevax ACWY.
  Interventions: Biological: Meningococcal vaccine GSK134612

INTERVENTIONS:
Biological: Meningococcal vaccine GSK134612 — One dose administered intramuscularly (IM) in the deltoid of the non-dominant arm

SUMMARY:
The purpose of this study is to evaluate the long-term antibody persistence 6, 7, 8, 9 and 10 years after receiving a primary vaccination of meningococcal conjugate vaccine MenACWY-TT versus Meningitec™ or Mencevax™ ACWY, and the safety and immunogenicity of a booster dose of MenACWY-TT administered 10 years after the primary vaccination. All subjects received a primary vaccination at 1 to 10 years of age in study 108658 (NCT00427908). No new subjects will be enrolled in this booster study.

DETAILED DESCRIPTION:
The study aims to evaluate the antibody persistence post primary vaccination with active control, safety and immunogenicity of a booster dose uncontrolled post primary vaccination during different phases:

Persistence phase: Long-term persistence 6, 7, 8, 9 and 10 years after primary vaccination with MenACWY-TT or Meningitec or Mencevax ACWY, in study MenACWY-TT-027.

Booster phase: One month post booster vaccination with MenACWY-TT vaccine ten years after primary vaccination.

The subjects in this study will be allocated to the same groups as in the vaccination study MenACWY-TT-027 (NCT00427908).

ELIGIBILITY:
Inclusion Criteria:

* Subjects and/or subjects' parent(s)/Legally Acceptable Representative(s) (LARs) who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* A male or female who has received a primary vaccination with the MenACWY-TT, Meningitec or Mencevax ACWY vaccines in study MenACWY-TT-027 (NCT00427908).
* In alignment with local laws and regulations, written informed consent obtained from parents/LAR(s) of the subject and written informed assent obtained from the subject if the subject is less than 15 years of age, or written informed consent obtained from the subject if the subject has achieved the 15th birthday. The subjects ≥15 years of age at the time of enrollment will sign the informed consent form, even if the parent/ LAR previously signed the ICF before the subject reached the legal age of consent.
* Healthy subjects as established by medical history and history-directed physical examination before entering into the study.

All subjects must satisfy the following additional criteria prior to entry of the booster phase:

* Female subjects of non-childbearing potential may be enrolled in the study.

  * Non-childbearing potential is defined as pre-menarche, hysterectomy or bilateral ovariectomy.
* Male subjects able to father children and female subjects of childbearing potential (including females who have had tubal ligation) and at risk of pregnancy may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination (for females only), and
  * has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination.

Exclusion Criteria:

* Child in care.
* Previous vaccination with meningococcal polysaccharide or conjugate vaccine outside of study MenACWY-TT-027.

Note: Subjects who were revaccinated with a monovalent MenC conjugate vaccine because of suboptimal response during the persistence phase of the MenACWY-TT-027 study (i.e. MenACWY-TT-028, -029, -030, -031 and -032) are allowed to participate as they will be followed for the persistence of MenA, MenW-135 and MenY.

* History of meningococcal disease due to serogroup A, C, W-135 or Y.
* Previous vaccination with meningococcal B vaccine.
* Any confirmed or suspected immunosuppressive or immunodeficient condition (congenital or secondary), including Human Immunodeficiency Virus (HIV) infection, based on medical history and physical examination (no laboratory testing required).
* Family history of congenital or hereditary immunodeficiency.
* Major congenital defects or serious chronic illness.
* History of chronic alcohol consumption and/or drug abuse.
* Subjects who withdrew consent to be contacted for follow-up studies.

Additional exclusion criteria for booster phase at Month 126 study entry (to be checked at Month 126) for all subjects:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine within 30 days preceding the booster dose of study vaccine, or planned use during the follow-up period.
* Administration of a vaccine not foreseen by the study protocol in the period starting 30 days before the booster dose of study vaccine or planned administration within 30 days after vaccination, with the exception of a licensed inactivated influenza vaccine.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the booster vaccine dose . Inhaled and topical steroids are allowed.
* Administration of immunoglobulins and/or any blood products within the three months preceding the booster vaccination or planned administration during the follow-up period.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product .
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccines.
* History of any neurological disorders or seizures, including Guillain-Barré syndrome (GBS). History of a simple, single febrile seizure is permitted.
* Acute disease and/or fever at the time of vaccination.

  * Fever is defined as temperature ≥ 37.5°C for oral, axillary, tympanic, or ≥38.0°C for rectal route. The preferred route for recording temperature in this study will be oral.
  * Subjects with a minor illness (such as mild diarrhoea, mild upper respiratory infection) without fever may, be enrolled at the discretion of the investigator.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.
* Male subjects able to father children who are planning to discontinue contraceptive precautions.
* Subjects who are investigational site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or subjects who are Pfizer employees directly involved in the conduct of the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (9):
- Finland (9):
  - Espoo Vaccine Research Clinic, Espoo
  - South Helsinki Vaccine Research Clinic, Helsinki
  - Helsinki East Vaccine Research Clinic, Helsinki
  - Jarvenpaa Vaccine Research Clinic, Jarvenpaa
  - Tampereen yliopisto/ Oulun rokotetutkimusklinikka, Oulu
  - Tampereen yliopisto/ Porin rokotetutkimusklinikka, Pori
  - Tampere Vaccine Research Clinic, Tampere
  - Tampereen yliopisto/ Turun rokotetutkimusklinikka, Turku
  - Tampereen yliopisto/ Ita-Vantaan rokotetutkimusklinikka, Vantaa

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Vesikari T, Peyrani P, Webber C, Van Der Wielen M, Cheuvart B, De Schrevel N, Aris E, Cutler M, Li P, Perez JL. Ten-Year Antibody Persistence and Booster Response to MenACWY-TT Vaccine After Primary Vaccination at 1-10 Years of Age. Hum Vaccin Immunother. 2020 Jun 2;16(6):1280-1291. doi: 10.1080/21645515.2020.1746110. PMID 32598244
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=MENACWY-TT-100&StudyName=A%20Phase%20Iiib%2C%20Open%2C%20Multi-center%20Study%20To%20Evaluate%20The%20Long-term%20Antibody%20Persistence%20At%206%2C%207%2C%208%2C%209%20And%2010%20Years%20After%20The%20Administration%20Of%20One%20Dose%20Of%20The%20Meningococcal%20Conjugate%20Vaccine%20Menacwy-tt%20Versus%20One%20Dose%20Of%20Meningitec%28registered%29%20Vaccine%20Or%20One%20Dose%20Of%20The%20Meningococcal%20Polysaccharide%20Vaccine%20Mencevax%28registered%29%20Acwy%2C%20And%20To%20Evaluate%20The%20Safety%20And%20Immunogenicity%20Of%20A%20Booster%20Dose%20Of%20Menacwy-tt%20Vaccine%20Administered%2010%20Years%20After%20Primary%20Vaccination%20Of%201-10%20Year%20Old%20Subjects%20With%20Menacwy-tt%2C%20Meningitec%28registered%29%20Or%20Mencevax%28registered%29%20Acwy.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In this study, participants from the study MENACWY-TT-027 [NCT00427908] were followed up for assessment of persistence of immune response and safety. And those who consented received booster vaccination and were followed up for another 6 months.
Groups:
- MenACWY-TT Vaccine: Less Than (<) 2 Years: Persistence phase was followed up by booster phase. Persistence phase: Participants with <2 years of age, received a single 0.5 milliliter (mL) dose of meningococcal serogroups A, C, W 135, Y tetanus toxoid conjugate (MenACWY-TT) vaccine intramuscularly, as primary vaccination in study MENACWY-TT-027. Then, in this study (MENACWY-TT-100), they were evaluated for long-term persistence (of immune response and safety) for 5 years (6, 7, 8, 9 and 10 years post primary vaccination). Booster phase: Participants who provided consent, received a single 0.5 mL booster dose of MenACWY-TT vaccine intramuscularly in this study, 10 years post primary vaccination in MENACWY-TT-027, and were followed up for 6 months after booster vaccination.
- MenCCRM (Meningitec) Vaccine: Less Than 2 Years: Persistence phase was followed up by booster phase. Persistence phase: Participants with <2 years of age, received a single 0.5 mL dose of Meningitec vaccine intramuscularly, as primary vaccination in study MENACWY-TT-027. Then, in this study (MENACWY-TT-100) they were evaluated for long-term persistence (of immune response and safety) for 5 years (6, 7, 8, 9 and 10 years post primary vaccination). Booster phase: Participants who provided consent, received a single 0.5 mL booster dose of MenACWY-TT vaccine intramuscularly in this study, 10 years post primary vaccination in MENACWY-TT-027, and were followed up for 6 months after booster vaccination.
- MenACWY-TT Vaccine: Greater Than or Equal to (>=) 2 Years: Persistence phase was followed up by booster phase. Persistence phase: Participants with >=2 years of age, received a single 0.5 mL dose of MenACWY-TT vaccine intramuscularly, as primary vaccination in study MENACWY-TT-027. Then, in this study (MENACWY-TT-100) they were evaluated for long-term persistence (of immune response and safety) for 5 years (6, 7, 8, 9 and 10 years post primary vaccination). Booster phase: Participants who provided consent, received a single 0.5 mL booster dose of MenACWY-TT vaccine intramuscularly in this study, 10 years post primary vaccination in MENACWY-TT-027, and were followed up for 6 months after booster vaccination.
- MenPS (Mencevax ACWY) Vaccine: Less Than 2 Years: Persistence phase was followed up by booster phase. Persistence phase: Participants with <2 years of age, received a single 0.5 mL dose of MencevaxACWY vaccine intramuscularly, as primary vaccination in study MENACWY-TT-027. Then, in this study (MENACWY-TT-100) they were evaluated for long term persistence (of immune response and safety) for 5 years (6, 7, 8, 9 and 10 years post primary vaccination). Booster phase: Participants who provided consent, received a single 0.5 mL booster dose of MenACWY-TT vaccine intramuscularly in this study, 10 years post primary vaccination in MENACWY-TT-027, and were followed up for 6 months after booster vaccination.
Period: Persistence Phase (5 Years)
Arm/Group | MenACWY-TT Vaccine: Less Than (<) 2 Years | MenCCRM (Meningitec) Vaccine: Less Than 2 Years | MenACWY-TT Vaccine: Greater Than or Equal to (>=) 2 Years | MenPS (Mencevax ACWY) Vaccine: Less Than 2 Years
Started | 76 | 23 | 115 | 29
Completed | 47 | 10 | 71 | 17
Not Completed | 29 | 13 | 44 | 12
Not completed — Lost to Follow-up | 2 | 1 | 5 | 2
Not completed — Migrated/moved from study area | 2 | 0 | 4 | 0
Not completed — Withdrawal by Subject | 4 | 5 | 18 | 4
Not completed — Eligibility criteria not fulfilled | 0 | 0 | 3 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Missed at least 1 persistence visit | 21 | 7 | 13 | 5
Period: Booster Phase (6 Months)
Arm/Group | MenACWY-TT Vaccine: Less Than (<) 2 Years | MenCCRM (Meningitec) Vaccine: Less Than 2 Years | MenACWY-TT Vaccine: Greater Than or Equal to (>=) 2 Years | MenPS (Mencevax ACWY) Vaccine: Less Than 2 Years
Started | 67 (Eligible participants from persistence phase who provided consent to get enrolled in booster phase.) | 16 (Eligible participants from persistence phase who provided consent to get enrolled in booster phase.) | 77 (Eligible participants from persistence phase who provided consent to get enrolled in booster phase.) | 21 (Eligible participants from persistence phase who provided consent to get enrolled in booster phase.)
Completed | 67 | 16 | 77 | 21
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all the participants enrolled in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | MenACWY-TT Vaccine: Less Than (<) 2 Years | MenCCRM (Meningitec) Vaccine: Less Than 2 Years | MenACWY-TT Vaccine: Greater Than or Equal to (>=) 2 Years | MenPS (Mencevax ACWY) Vaccine: Less Than 2 Years | Total
Number analyzed (Participants) | 76 | 23 | 115 | 29 | 243
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.2 (0.7) | 8.2 (0.7) | 12.5 (2.6) | 12.1 (2.9) | 10.7 (3.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 12 | 56 | 14 | 122
  Male | 36 | 11 | 59 | 15 | 121
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 76 | 23 | 115 | 29 | 243
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White - Arabic/North African heritage | 0 | 0 | 1 | 0 | 1
  White - Caucasian/European heritage | 75 | 22 | 113 | 28 | 238
  Other | 1 | 1 | 1 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Persistence Phase: Percentage of Participants With Serum Bactericidal Assay Using Rabbit Complement (rSBA) Titers >=1:8 and >=1:128 For Each of the 4 Serogroups After 6 Years of Primary Vaccination
Description: Serogroups included Neisseria meningitidis serogroup A (MenA), Neisseria meningitidis serogroup C (MenC), Neisseria meningitidis serogroup W-135 (MenW-135) and Neisseria meningitidis serogroup Y (MenY).
Time Frame: 6 years after primary vaccination (Year 1 of study MENACWY-TT-100)
Population: All eligible participants who received primary vaccination with MenACWY-TT, Meningitec, or Mencevax ACWY during study MenACWY-TT-027 and had available assay results for at least 1 tested antigen. Here, "Overall Number of Participants Analyzed" (N) signifies number of participants evaluable for this measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MenACWY-TT Vaccine: Less Than (<) 2 Years | MenCCRM (Meningitec) Vaccine: Less Than 2 Years | MenACWY-TT Vaccine: Greater Than or Equal to (>=) 2 Years | MenPS (Mencevax ACWY) Vaccine: Less Than 2 Years
Number analyzed (Participants) | 54 | 16 | 98 | 24
percentage of participants
  rSBA-MenA: >=1:8 | 51.9 [37.8 to 65.7] | 18.8 [4.0 to 45.6] | 79.6 [70.3 to 87.1] | 12.5 [2.7 to 32.4]
  rSBA-MenC: >=1:8 | 77.8 [64.4 to 88.0] | 75.0 [47.6 to 92.7] | 82.7 [73.7 to 89.6] | 79.2 [57.8 to 92.9]
  rSBA-MenW-135: >=1:8 | 33.3 [21.1 to 47.5] | 12.5 [1.6 to 38.3] | 73.5 [63.6 to 81.9] | 12.5 [2.7 to 32.4]
  rSBA-MenY: >=1:8 | 38.9 [25.9 to 53.1] | 37.5 [15.2 to 64.6] | 71.4 [61.4 to 80.1] | 20.8 [7.1 to 42.2]
  rSBA-MenA: >=1:28 | 16.7 [7.9 to 29.3] | 6.3 [0.2 to 30.2] | 55.1 [44.7 to 65.2] | 8.3 [1.0 to 27.0]
  rSBA-MenC: >=1:28 | 70.4 [56.4 to 82.0] | 56.3 [29.9 to 80.2] | 68.4 [58.2 to 77.4] | 62.5 [40.6 to 81.2]
  rSBA-MenW-135: >=1:28 | 29.6 [18.0 to 43.6] | 6.3 [0.2 to 30.2] | 73.5 [63.6 to 81.9] | 12.5 [2.7 to 32.4]
  rSBA-MenY: >=1:28 | 33.3 [21.1 to 47.5] | 31.3 [11.0 to 58.7] | 65.3 [55.0 to 74.6] | 20.8 [7.1 to 42.2]

2. Primary Outcome: Persistence Phase: Percentage of Participants With rSBA Titers >= 1:8 and >=1:128 For Each of the 4 Serogroups After 7 Years of Primary Vaccination
Description: Serogroups included MenA, MenC, MenW-135 and MenY.
Time Frame: 7 years after primary vaccination (Year 2 of study MENACWY-TT-100)
Population: All eligible participants who received primary vaccination with MenACWY-TT, Meningitec or Mencevax ACWY in Study MenACWY-TT-027, had available assay results for at least 1 tested antigen. "N": number of participants evaluable for this measure. "Number analyzed": participants analyzed for specified serogroup titers cut off.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MenACWY-TT Vaccine: Less Than (<) 2 Years | MenCCRM (Meningitec) Vaccine: Less Than 2 Years | MenACWY-TT Vaccine: Greater Than or Equal to (>=) 2 Years | MenPS (Mencevax ACWY) Vaccine: Less Than 2 Years
Number analyzed (Participants) | 60 | 21 | 104 | 27
percentage of participants
  rSBA-MenA: >=1:8 | 58.3 [44.9 to 70.9] | 9.5 [1.2 to 30.4] | 74.0 [64.5 to 82.1] | 18.5 [6.3 to 38.1]
  rSBA-MenC: >=1:8: number analyzed (Participants) | 60 | 21 | 101 | 27
  rSBA-MenC: >=1:8 | 78.3 [65.8 to 87.9] | 71.4 [47.8 to 88.7] | 84.2 [75.6 to 90.7] | 81.5 [61.9 to 93.7]
  rSBA-MenW-135: >=1:8: number analyzed (Participants) | 60 | 21 | 102 | 27
  rSBA-MenW-135: >=1:8 | 26.7 [16.1 to 39.7] | 9.5 [1.2 to 30.4] | 73.5 [63.9 to 81.8] | 11.1 [2.4 to 29.2]
  rSBA-MenY: >=1:8: number analyzed (Participants) | 60 | 21 | 102 | 27
  rSBA-MenY: >=1:8 | 35.0 [23.1 to 48.4] | 28.6 [11.3 to 52.2] | 75.5 [66.0 to 83.5] | 14.8 [4.2 to 33.7]
  rSBA-MenA: >=1:28 | 21.7 [12.1 to 34.2] | 9.5 [1.2 to 30.4] | 44.2 [34.5 to 54.3] | 11.1 [2.4 to 29.2]
  rSBA-MenC: >=1:28: number analyzed (Participants) | 60 | 21 | 101 | 27
  rSBA-MenC: >=1:28 | 61.7 [48.2 to 73.9] | 52.4 [29.8 to 74.3] | 61.4 [51.2 to 70.9] | 66.7 [46.0 to 83.5]
  rSBA-MenW-135: >=1:28: number analyzed (Participants) | 60 | 21 | 102 | 27
  rSBA-MenW-135: >=1:28 | 23.3 [13.4 to 36.0] | 9.5 [1.2 to 30.4] | 69.6 [59.7 to 78.3] | 7.4 [0.9 to 24.3]
  rSBA-MenY: >=1:28: number analyzed (Participants) | 60 | 21 | 102 | 27
  rSBA-MenY: >=1:28 | 33.3 [21.7 to 46.7] | 28.6 [11.3 to 52.2] | 69.6 [59.7 to 78.3] | 14.8 [4.2 to 33.7]

3. Primary Outcome: Persistence Phase: Percentage of Participants With rSBA Titers >= 1:8 and >=1:128 For Each of the 4 Serogroups After 8 Years of Primary Vaccination
Description: Serogroups included MenA, MenC, MenW-135 and MenY.
Time Frame: 8 years after primary vaccination (Year 3 of study MENACWY-TT-100)
Population: All eligible participants who received primary vaccination with MenACWY-TT, Meningitec or Mencevax ACWY in Study MenACWY-TT-027 and had available assay results for at least 1 tested antigen. "N": number of participants evaluable for this measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MenACWY-TT Vaccine: Less Than (<) 2 Years | MenCCRM (Meningitec) Vaccine: Less Than 2 Years | MenACWY-TT Vaccine: Greater Than or Equal to (>=) 2 Years | MenPS (Mencevax ACWY) Vaccine: Less Than 2 Years
Number analyzed (Participants) | 65 | 22 | 100 | 25
percentage of participants
  rSBA-MenA: >=1:8 | 47.7 [35.1 to 60.5] | 4.5 [0.1 to 22.8] | 70.0 [60.0 to 78.8] | 24.0 [9.4 to 45.1]
  rSBA-MenC: >=1:8 | 78.5 [66.5 to 87.7] | 77.3 [54.6 to 92.2] | 85.0 [76.5 to 91.4] | 88.0 [68.8 to 97.5]
  rSBA-MenW-135: >=1:8 | 29.2 [18.6 to 41.8] | 13.6 [2.9 to 34.9] | 76.0 [66.4 to 84.0] | 20.0 [6.8 to 40.7]
  rSBA-MenY: >=1:8 | 40.0 [28.0 to 52.9] | 40.9 [20.7 to 63.6] | 79.0 [69.7 to 86.5] | 24.0 [9.4 to 45.1]
  rSBA-MenA: >=1:28 | 23.1 [13.5 to 35.2] | 4.5 [0.1 to 22.8] | 45.0 [35.0 to 55.3] | 12.0 [2.5 to 31.2]
  rSBA-MenC: >=1:28 | 64.6 [51.8 to 76.1] | 50.0 [28.2 to 71.8] | 61.0 [50.7 to 70.6] | 64.0 [42.5 to 82.0]
  rSBA-MenW-135: >=1:28 | 27.7 [17.3 to 40.2] | 9.1 [1.1 to 29.2] | 76.0 [66.4 to 84.0] | 20.0 [6.8 to 40.7]
  rSBA-MenY: >=1:28 | 38.5 [26.7 to 51.4] | 40.9 [20.7 to 63.6] | 73.0 [63.2 to 81.4] | 20.0 [6.8 to 40.7]

4. Primary Outcome: Persistence Phase: Percentage of Participants With rSBA Titers >= 1:8 and >=1:128 For Each of the 4 Serogroups After 9 Years of Primary Vaccination
Description: Serogroups included MenA, MenC, MenW-135 and MenY.
Time Frame: 9 years after primary vaccination (Year 4 of study MENACWY-TT-100)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MenACWY-TT Vaccine: Less Than (<) 2 Years | MenCCRM (Meningitec) Vaccine: Less Than 2 Years | MenACWY-TT Vaccine: Greater Than or Equal to (>=) 2 Years | MenPS (Mencevax ACWY) Vaccine: Less Than 2 Years
Number analyzed (Participants) | 64 | 21 | 93 | 25
percentage of participants
  rSBA-MenA >=1:8 | 67.2 [54.3 to 78.4] | 4.8 [0.1 to 23.8] | 79.6 [69.9 to 87.2] | 24.0 [9.4 to 45.1]
  rSBA-MenC >=1:8 | 81.3 [69.5 to 89.9] | 85.7 [63.7 to 97.0] | 86.0 [77.3 to 92.3] | 84.0 [63.9 to 95.5]
  rSBA-MenW-135 >=1:8: number analyzed (Participants) | 64 | 21 | 92 | 25
  rSBA-MenW-135 >=1:8 | 32.8 [21.6 to 45.7] | 9.5 [1.2 to 30.4] | 76.1 [66.1 to 84.4] | 16.0 [4.5 to 36.1]
  rSBA-MenY >=1:8 | 42.2 [29.9 to 55.2] | 47.6 [25.7 to 70.2] | 66.7 [56.1 to 76.1] | 20.0 [6.8 to 40.7]
  rSBA-MenA >=1:28 | 31.3 [20.2 to 44.1] | 4.8 [0.1 to 23.8] | 57.0 [46.3 to 67.2] | 16.0 [4.5 to 36.1]
  rSBA-MenC >=1:28 | 65.6 [52.7 to 77.1] | 57.1 [34.0 to 78.2] | 64.5 [53.9 to 74.2] | 68.0 [46.5 to 85.1]
  rSBA-MenW-135 >=1:28: number analyzed (Participants) | 64 | 21 | 92 | 25
  rSBA-MenW-135 >=1:28 | 26.6 [16.3 to 39.1] | 9.5 [1.2 to 30.4] | 71.7 [61.4 to 80.6] | 16.0 [4.5 to 36.1]
  rSBA-MenY >=1:28 | 34.4 [22.9 to 47.3] | 38.1 [18.1 to 61.6] | 58.1 [47.4 to 68.2] | 16.0 [4.5 to 36.1]

5. Primary Outcome: Persistence Phase: Percentage of Participants With rSBA Titers >= 1:8 and >=1:128 For Each of the 4 Serogroups After 10 Years of Primary Vaccination
Description: Serogroups included MenA, MenC, MenW-135 and MenY.
Time Frame: 10 years after primary vaccination (Year 4 of study MENACWY-TT-100)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MenACWY-TT Vaccine: Less Than (<) 2 Years | MenCCRM (Meningitec) Vaccine: Less Than 2 Years | MenACWY-TT Vaccine: Greater Than or Equal to (>=) 2 Years | MenPS (Mencevax ACWY) Vaccine: Less Than 2 Years
Number analyzed (Participants) | 64 | 17 | 82 | 21
percentage of participants
  rSBA-MenA >=1:8: number analyzed (Participants) | 64 | 17 | 81 | 21
  rSBA-MenA >=1:8 | 65.6 [52.7 to 77.1] | 17.6 [3.8 to 43.4] | 88.9 [80.0 to 94.8] | 28.6 [11.3 to 52.2]
  rSBA-MenC >=1:8 | 82.8 [71.3 to 91.1] | 88.2 [63.6 to 98.5] | 84.1 [74.4 to 91.3] | 81.0 [58.1 to 94.6]
  rSBA-MenW-135 >=1:8 | 31.3 [20.2 to 44.1] | 0.0 [0.0 to 19.5] | 67.1 [55.8 to 77.1] | 23.8 [8.2 to 47.2]
  rSBA-MenY >=1:8 | 43.8 [31.4 to 56.7] | 35.3 [14.2 to 61.7] | 65.9 [54.6 to 76.0] | 23.8 [8.2 to 47.2]
  rSBA-MenA >=1:28: number analyzed (Participants) | 64 | 17 | 81 | 21
  rSBA-MenA >=1:28 | 26.6 [16.3 to 39.1] | 5.9 [0.1 to 28.7] | 49.4 [38.1 to 60.7] | 14.3 [3.0 to 36.3]
  rSBA-MenC >=1:28 | 64.1 [51.1 to 75.7] | 58.8 [32.9 to 81.6] | 65.9 [54.6 to 76.0] | 66.7 [43.0 to 85.4]
  rSBA-MenW-135 >=1:28 | 28.1 [17.6 to 40.8] | 0.0 [0.0 to 19.5] | 65.9 [54.6 to 76.0] | 23.8 [8.2 to 47.2]
  rSBA-MenY >=1:28 | 35.9 [24.3 to 48.9] | 29.4 [10.3 to 56.0] | 59.8 [48.3 to 70.4] | 19.0 [5.4 to 41.9]

6. Primary Outcome: Persistence Phase: Geometric Mean Titers as Measured by rSBA for Each of the 4 Serogroups After 6 Years of Primary Vaccination
Description: Serogroups included MenA, MenC, MenW-135 and MenY.
Time Frame: 6 Years after primary vaccination (Year 1 of study MENACWY-TT-100)
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | MenACWY-TT Vaccine: Less Than (<) 2 Years | MenCCRM (Meningitec) Vaccine: Less Than 2 Years | MenACWY-TT Vaccine: Greater Than or Equal to (>=) 2 Years | MenPS (Mencevax ACWY) Vaccine: Less Than 2 Years
Number analyzed (Participants) | 54 | 16 | 98 | 24
titers
  rSBA-MenA | 16.0 [9.8 to 26.1] | 5.9 [3.1 to 11.3] | 107.3 [66.0 to 174.3] | 5.8 [3.5 to 9.6]
  rSBA-MenC | 161.3 [84.7 to 307.1] | 103.1 [31.9 to 333.3] | 192.9 [121.0 to 307.5] | 98.7 [42.2 to 230.7]
  rSBA-MenW-135 | 18.0 [9.8 to 32.9] | 6.2 [3.1 to 12.3] | 265.2 [154.9 to 454.1] | 7.6 [3.7 to 15.6]
  rSBA-MenY | 21.5 [11.5 to 40.1] | 21.7 [5.9 to 79.0] | 136.4 [82.6 to 225.3] | 11.6 [4.7 to 28.7]

7. Primary Outcome: Persistence Phase: Geometric Mean Titers as Measured by rSBA for Each of the 4 Serogroups After 7 Years of Primary Vaccination
Description: Serogroups included MenA, MenC, MenW-135 and MenY.
Time Frame: 7 years after primary vaccination (Year 2 of study MENACWY-TT-100)
Population: All eligible participants who received primary vaccination with MenACWY-TT, Meningitec or Mencevax ACWY in Study MenACWY-TT-027, had available assay results for at least 1 tested antigen. "N": number of participants evaluable for this measure. "Number analyzed": participants analyzed for specified serogroup.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | MenACWY-TT Vaccine: Less Than (<) 2 Years | MenCCRM (Meningitec) Vaccine: Less Than 2 Years | MenACWY-TT Vaccine: Greater Than or Equal to (>=) 2 Years | MenPS (Mencevax ACWY) Vaccine: Less Than 2 Years
Number analyzed (Participants) | 60 | 21 | 104 | 27
titers
  rSBA-MenA | 20.4 [12.1 to 34.4] | 6.1 [3.3 to 11.4] | 65.3 [40.5 to 105.4] | 7.4 [4.0 to 13.8]
  rSBA-MenC: number analyzed (Participants) | 60 | 21 | 101 | 27
  rSBA-MenC | 104.0 [58.0 to 186.3] | 54.3 [18.5 to 158.9] | 139.0 [87.8 to 220.0] | 101.6 [42.1 to 245.0]
  rSBA-MenW-135: number analyzed (Participants) | 60 | 21 | 102 | 27
  rSBA-MenW-135 | 13.0 [7.6 to 22.3] | 6.8 [3.0 to 15.3] | 206.0 [120.9 to 350.9] | 6.3 [3.7 to 10.9]
  rSBA-MenY: number analyzed (Participants) | 60 | 21 | 102 | 27
  rSBA-MenY | 19.9 [11.0 to 36.1] | 18.3 [5.8 to 57.6] | 152.7 [96.1 to 242.6] | 8.2 [4.1 to 16.5]

8. Primary Outcome: Persistence Phase: Geometric Mean Titers as Measured by rSBA for Each of the 4 Serogroups After 8 Years of Primary Vaccination
Description: Serogroups included MenA, MenC, MenW-135 and MenY.
Time Frame: 8 years after primary vaccination (Year 3 of study MENACWY-TT-100)
Population: All eligible participants who received primary vaccination with MenACWY-TT, Meningitec or Mencevax ACWY in Study MenACWY-TT-027, had available assay results for at least 1 tested antigen. "N": number of participants evaluable for this measure.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | MenACWY-TT Vaccine: Less Than (<) 2 Years | MenCCRM (Meningitec) Vaccine: Less Than 2 Years | MenACWY-TT Vaccine: Greater Than or Equal to (>=) 2 Years | MenPS (Mencevax ACWY) Vaccine: Less Than 2 Years
Number analyzed (Participants) | 65 | 22 | 100 | 25
titers
  rSBA-MenA | 15.8 [9.8 to 25.6] | 4.8 [3.3 to 7.2] | 51.3 [31.5 to 83.4] | 7.8 [4.2 to 14.3]
  rSBA-MenC | 110.2 [65.9 to 184.3] | 64.0 [26.0 to 157.4] | 140.1 [91.3 to 214.9] | 121.1 [52.2 to 281.1]
  rSBA-MenW-135 | 15.3 [9.0 to 26.3] | 6.4 [3.3 to 12.4] | 252.5 [154.3 to 413.2] | 11.8 [4.7 to 29.8]
  rSBA-MenY | 26.1 [14.4 to 47.5] | 33.0 [9.8 to 111.0] | 181.0 [115.0 to 284.9] | 10.9 [4.8 to 24.6]

9. Primary Outcome: Persistence Phase: Geometric Mean Titers as Measured by rSBA for Each of the 4 Serogroups After 9 Years of Primary Vaccination
Description: Serogroups included MenA, MenC, MenW-135 and MenY.
Time Frame: 9 years after primary vaccination (Year 4 of study MENACWY-TT-100)
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | MenACWY-TT Vaccine: Less Than (<) 2 Years | MenCCRM (Meningitec) Vaccine: Less Than 2 Years | MenACWY-TT Vaccine: Greater Than or Equal to (>=) 2 Years | MenPS (Mencevax ACWY) Vaccine: Less Than 2 Years
Number analyzed (Participants) | 64 | 21 | 93 | 25
titers
  rSBA-MenA | 28.4 [16.5 to 48.9] | 5.2 [3.0 to 9.0] | 118.8 [71.1 to 198.6] | 10.9 [4.5 to 26.2]
  rSBA-MenC | 166.0 [92.3 to 298.7] | 92.0 [32.7 to 259.1] | 176.4 [106.8 to 291.3] | 164.3 [66.5 to 405.8]
  rSBA-MenW-135: number analyzed (Participants) | 64 | 21 | 92 | 25
  rSBA-MenW-135 | 17.3 [9.7 to 30.8] | 6.6 [3.2 to 13.6] | 274.0 [155.8 to 481.7] | 9.7 [4.0 to 23.3]
  rSBA-MenY | 23.1 [13.0 to 41.2] | 32.0 [10.6 to 96.3] | 106.2 [61.5 to 183.4] | 10.0 [4.4 to 22.9]

10. Primary Outcome: Persistence Phase: Geometric Mean Titers as Measured by rSBA for Each of the 4 Serogroups After 10 Years of Primary Vaccination
Description: Serogroups included MenA, MenC, MenW-135 and MenY.
Time Frame: 10 years after primary vaccination (Year 5 of study MENACWY-TT-100)
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | MenACWY-TT Vaccine: Less Than (<) 2 Years | MenCCRM (Meningitec) Vaccine: Less Than 2 Years | MenACWY-TT Vaccine: Greater Than or Equal to (>=) 2 Years | MenPS (Mencevax ACWY) Vaccine: Less Than 2 Years
Number analyzed (Participants) | 64 | 17 | 82 | 21
titers
  rSBA-MenA: number analyzed (Participants) | 64 | 17 | 81 | 21
  rSBA-MenA | 29.3 [16.8 to 51.3] | 5.8 [3.2 to 10.6] | 106.0 [63.7 to 176.4] | 9.1 [4.0 to 20.7]
  rSBA-MenC | 132.2 [74.5 to 234.6] | 81.7 [29.2 to 229.2] | 175.0 [104.7 to 292.4] | 105.0 [37.2 to 296.4]
  rSBA-MenW-135 | 16.7 [9.5 to 29.3] | 4.0 [NA to NA] — The confidence interval was not estimable due to the lack of variability of antibody titer. | 187.2 [101.0 to 347.1] | 14.0 [4.8 to 41.2]
  rSBA-MenY | 25.8 [14.0 to 47.3] | 22.2 [5.8 to 84.2] | 90.5 [51.5 to 159.2] | 12.7 [4.2 to 38.1]

11. Secondary Outcome: Persistence Phase: Percentage of Participants With Serum Bactericidal Assay Using Human Complement (hSBA) Titers >=1:4 and >=1:8 for Each of the 4 Serogroups After 6, 7, 8, 9 and 10 Years of Primary Vaccination
Description: Serogroups included MenA, MenC, MenW-135 and MenY.
Time Frame: 6, 7, 8, 9 and 10 years after primary vaccination (Year 1, 2, 3, 4 and 5 of study MENACWY-TT-100)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MenACWY-TT Vaccine: Less Than (<) 2 Years | MenCCRM (Meningitec) Vaccine: Less Than 2 Years | MenACWY-TT Vaccine: Greater Than or Equal to (>=) 2 Years | MenPS (Mencevax ACWY) Vaccine: Less Than 2 Years
Number analyzed (Participants) | 64 | 22 | 100 | 27
percentage of participants
  Year 1 of study MENACWY-TT-100: hSBA-MenA >=1:4: number analyzed (Participants) | 44 | 14 | 90 | 21
  Year 1 of study MENACWY-TT-100: hSBA-MenA >=1:4 | 34.1 [20.5 to 49.9] | 28.6 [8.4 to 58.1] | 42.2 [31.9 to 53.1] | 42.9 [21.8 to 66.0]
  Year 2 of study MENACWY-TT-10: hSBA-MenA >=1:4: number analyzed (Participants) | 60 | 21 | 99 | 26
  Year 2 of study MENACWY-TT-10: hSBA-MenA >=1:4 | 26.7 [16.1 to 39.7] | 14.3 [3.0 to 36.3] | 26.3 [17.9 to 36.1] | 26.9 [11.6 to 47.8]
  Year 3 of study MENACWY-TT-10: hSBA-MenA >=1:4: number analyzed (Participants) | 64 | 22 | 97 | 25
  Year 3 of study MENACWY-TT-10: hSBA-MenA >=1:4 | 32.8 [21.6 to 45.7] | 27.3 [10.7 to 50.2] | 28.9 [20.1 to 39.0] | 40.0 [21.1 to 61.3]
  Year 4 of study MENACWY-TT-10: hSBA-MenA >=1:4: number analyzed (Participants) | 63 | 20 | 86 | 23
  Year 4 of study MENACWY-TT-10: hSBA-MenA >=1:4 | 39.7 [27.6 to 52.8] | 30.0 [11.9 to 54.3] | 43.0 [32.4 to 54.2] | 30.4 [13.2 to 52.9]
  Year 5 of study MENACWY-TT-10: hSBA-MenA >=1:4: number analyzed (Participants) | 61 | 16 | 69 | 21
  Year 5 of study MENACWY-TT-10: hSBA-MenA >=1:4 | 31.1 [19.9 to 44.3] | 25.0 [7.3 to 52.4] | 34.8 [23.7 to 47.2] | 33.3 [14.6 to 57.0]
  Year 1 of study MENACWY-TT-10: hSBA-MenC >=1:4: number analyzed (Participants) | 53 | 16 | 97 | 24
  Year 1 of study MENACWY-TT-10: hSBA-MenC >=1:4 | 92.5 [81.8 to 97.9] | 93.8 [69.8 to 99.8] | 93.8 [87.0 to 97.7] | 100.0 [85.8 to 100.0]
  Year 2 of study MENACWY-TT-10: hSBA-MenC >=1:4: number analyzed (Participants) | 59 | 20 | 96 | 26
  Year 2 of study MENACWY-TT-10: hSBA-MenC >=1:4 | 89.8 [79.2 to 96.2] | 100.0 [83.2 to 100.0] | 88.5 [80.4 to 94.1] | 92.3 [74.9 to 99.1]
  Year 3 of study MENACWY-TT-10: hSBA-MenC >=1:4: number analyzed (Participants) | 64 | 22 | 96 | 25
  Year 3 of study MENACWY-TT-10: hSBA-MenC >=1:4 | 92.2 [82.7 to 97.4] | 95.5 [77.2 to 99.9] | 89.6 [81.7 to 94.9] | 96.0 [79.6 to 99.9]
  Year 4 of study MENACWY-TT-10: hSBA-MenC >=1:4: number analyzed (Participants) | 63 | 20 | 90 | 24
  Year 4 of study MENACWY-TT-10: hSBA-MenC >=1:4 | 90.5 [80.4 to 96.4] | 95.0 [75.1 to 99.9] | 86.7 [77.9 to 92.9] | 91.7 [73.0 to 99.0]
  Year 5 of study MENACWY-TT-10: hSBA-MenC >=1:4: number analyzed (Participants) | 62 | 16 | 79 | 21
  Year 5 of study MENACWY-TT-10: hSBA-MenC >=1:4 | 91.9 [82.2 to 97.3] | 93.8 [69.8 to 99.8] | 91.1 [82.6 to 96.4] | 100.0 [83.9 to 100.0]
  Year 1 of study MENACWY-TT-10: hSBA-MenW-135>=1:4: number analyzed (Participants) | 47 | 15 | 92 | 23
  Year 1 of study MENACWY-TT-10: hSBA-MenW-135>=1:4 | 70.2 [55.1 to 82.7] | 13.3 [1.7 to 40.5] | 81.5 [72.1 to 88.9] | 30.4 [13.2 to 52.9]
  Year 2 of study MENACWY-TT-10: hSBA-MenW-135>=1:4: number analyzed (Participants) | 58 | 20 | 98 | 27
  Year 2 of study MENACWY-TT-10: hSBA-MenW-135>=1:4 | 60.3 [46.6 to 73.0] | 20.0 [5.7 to 43.7] | 79.6 [70.3 to 87.1] | 18.5 [6.3 to 38.1]
  Year 3 of study MENACWY-TT-10: hSBA-MenW-135>=1:4: number analyzed (Participants) | 64 | 21 | 94 | 25
  Year 3 of study MENACWY-TT-10: hSBA-MenW-135>=1:4 | 39.1 [27.1 to 52.1] | 19.0 [5.4 to 41.9] | 56.4 [45.8 to 66.6] | 12.0 [2.5 to 31.2]
  Year 4 of study MENACWY-TT-10: hSBA-MenW-135>=1:4: number analyzed (Participants) | 58 | 16 | 79 | 21
  Year 4 of study MENACWY-TT-10: hSBA-MenW-135>=1:4 | 44.8 [31.7 to 58.5] | 18.8 [4.0 to 45.6] | 68.4 [56.9 to 78.4] | 9.5 [1.2 to 30.4]
  Year 5 of study MENACWY-TT-10: hSBA-MenW-135>=1:4: number analyzed (Participants) | 54 | 14 | 67 | 19
  Year 5 of study MENACWY-TT-10: hSBA-MenW-135>=1:4 | 44.4 [30.9 to 58.6] | 21.4 [4.7 to 50.8] | 61.2 [48.5 to 72.9] | 26.3 [9.1 to 51.2]
  Year 1 of study MENACWY-TT-10: hSBA-MenY>=1:4: number analyzed (Participants) | 41 | 14 | 89 | 24
  Year 1 of study MENACWY-TT-10: hSBA-MenY>=1:4 | 31.7 [18.1 to 48.1] | 7.1 [0.2 to 33.9] | 65.2 [54.3 to 75.0] | 25.0 [9.8 to 46.7]
  Year 2 of study MENACWY-TT-10: hSBA-MenY>=1:4: number analyzed (Participants) | 56 | 21 | 100 | 27
  Year 2 of study MENACWY-TT-10: hSBA-MenY>=1:4 | 51.8 [38.0 to 65.3] | 33.3 [14.6 to 57.0] | 75.0 [65.3 to 83.1] | 40.7 [22.4 to 61.2]
  Year 3 of study MENACWY-TT-10: hSBA-MenY>=1:4: number analyzed (Participants) | 63 | 21 | 93 | 23
  Year 3 of study MENACWY-TT-10: hSBA-MenY>=1:4 | 50.8 [37.9 to 63.6] | 38.1 [18.1 to 61.6] | 72.0 [61.8 to 80.9] | 34.8 [16.4 to 57.3]
  Year 4 of study MENACWY-TT-10: hSBA-MenY>=1:4: number analyzed (Participants) | 61 | 19 | 84 | 22
  Year 4 of study MENACWY-TT-10: hSBA-MenY>=1:4 | 32.8 [21.3 to 46.0] | 26.3 [9.1 to 51.2] | 67.9 [56.8 to 77.6] | 27.3 [10.7 to 50.2]
  Year 5 of study MENACWY-TT-10: hSBA-MenY>=1:4: number analyzed (Participants) | 58 | 15 | 73 | 18
  Year 5 of study MENACWY-TT-10: hSBA-MenY>=1:4 | 41.4 [28.6 to 55.1] | 40.0 [16.3 to 67.7] | 72.6 [60.9 to 82.4] | 44.4 [21.5 to 69.2]
  Year 1 of study MENACWY-TT-10: hSBA-MenA>=1:8: number analyzed (Participants) | 44 | 14 | 90 | 21
  Year 1 of study MENACWY-TT-10: hSBA-MenA>=1:8 | 31.8 [18.6 to 47.6] | 28.6 [8.4 to 58.1] | 41.1 [30.8 to 52.0] | 33.3 [14.6 to 57.0]
  Year 2 of study MENACWY-TT-10: hSBA-MenA>=1:8: number analyzed (Participants) | 60 | 21 | 99 | 26
  Year 2 of study MENACWY-TT-10: hSBA-MenA>=1:8 | 25.0 [14.7 to 37.9] | 14.3 [3.0 to 36.3] | 26.3 [17.9 to 36.1] | 23.1 [9.0 to 43.6]
  Year 3 of study MENACWY-TT-10: hSBA-MenA>=1:8: number analyzed (Participants) | 64 | 22 | 97 | 25
  Year 3 of study MENACWY-TT-10: hSBA-MenA>=1:8 | 32.8 [21.6 to 45.7] | 27.3 [10.7 to 50.2] | 28.9 [20.1 to 39.0] | 36.0 [18.0 to 57.5]
  Year 4 of study MENACWY-TT-10: hSBA-MenA>=1:8: number analyzed (Participants) | 63 | 20 | 86 | 23
  Year 4 of study MENACWY-TT-10: hSBA-MenA>=1:8 | 30.2 [19.2 to 43.0] | 20.0 [5.7 to 43.7] | 43.0 [32.4 to 54.2] | 26.1 [10.2 to 48.4]
  Year 5 of study MENACWY-TT-10: hSBA-MenA>=1:8: number analyzed (Participants) | 61 | 16 | 69 | 21
  Year 5 of study MENACWY-TT-10: hSBA-MenA>=1:8 | 26.2 [15.8 to 39.1] | 18.8 [4.0 to 45.6] | 33.3 [22.4 to 45.7] | 28.6 [11.3 to 52.2]
  Year 1 of study MENACWY-TT-10: hSBA-MenC>=1:8: number analyzed (Participants) | 53 | 16 | 97 | 24
  Year 1 of study MENACWY-TT-10: hSBA-MenC>=1:8 | 92.5 [81.8 to 97.9] | 93.8 [69.8 to 99.8] | 93.8 [87.0 to 97.7] | 100.0 [85.8 to 100.0]
  Year 2 of study MENACWY-TT-10: hSBA-MenC>=1:8: number analyzed (Participants) | 59 | 20 | 96 | 26
  Year 2 of study MENACWY-TT-10: hSBA-MenC>=1:8 | 89.8 [79.2 to 96.2] | 100.0 [83.2 to 100.0] | 88.5 [80.4 to 94.1] | 92.3 [74.9 to 99.1]
  Year 3 of study MENACWY-TT-10: hSBA-MenC>=1:8: number analyzed (Participants) | 64 | 22 | 96 | 25
  Year 3 of study MENACWY-TT-10: hSBA-MenC>=1:8 | 92.2 [82.7 to 97.4] | 95.5 [77.2 to 99.9] | 89.6 [81.7 to 94.9] | 96.0 [79.6 to 99.9]
  Year 4 of study MENACWY-TT-10: hSBA-MenC>=1:8: number analyzed (Participants) | 63 | 20 | 90 | 24
  Year 4 of study MENACWY-TT-10: hSBA-MenC>=1:8 | 90.5 [80.4 to 96.4] | 95.0 [75.1 to 99.9] | 85.6 [76.6 to 92.1] | 91.7 [73.0 to 99.0]
  Year 5 of study MENACWY-TT-10: hSBA-MenC>=1:8: number analyzed (Participants) | 62 | 16 | 79 | 21
  Year 5 of study MENACWY-TT-10: hSBA-MenC>=1:8 | 91.9 [82.2 to 97.3] | 93.8 [69.8 to 99.8] | 91.1 [82.6 to 96.4] | 100.0 [83.9 to 100.0]
  Year 1 of study MENACWY-TT-10: hSBA-MenW-135 >=1:8: number analyzed (Participants) | 47 | 15 | 92 | 23
  Year 1 of study MENACWY-TT-10: hSBA-MenW-135 >=1:8 | 70.2 [55.1 to 82.7] | 13.3 [1.7 to 40.5] | 81.5 [72.1 to 88.9] | 30.4 [13.2 to 52.9]
  Year 2 of study MENACWY-TT-10: hSBA-MenW-135 >=1:8: number analyzed (Participants) | 58 | 20 | 98 | 27
  Year 2 of study MENACWY-TT-10: hSBA-MenW-135 >=1:8 | 60.3 [46.6 to 73.0] | 20.0 [5.7 to 43.7] | 79.6 [70.3 to 87.1] | 18.5 [6.3 to 38.1]
  Year 3 of study MENACWY-TT-10: hSBA-MenW-135 >=1:8: number analyzed (Participants) | 64 | 21 | 94 | 25
  Year 3 of study MENACWY-TT-10: hSBA-MenW-135 >=1:8 | 39.1 [27.1 to 52.1] | 19.0 [5.4 to 41.9] | 56.4 [45.8 to 66.6] | 12.0 [2.5 to 31.2]
  Year 4 of study MENACWY-TT-10: hSBA-MenW-135 >=1:8: number analyzed (Participants) | 58 | 16 | 79 | 21
  Year 4 of study MENACWY-TT-10: hSBA-MenW-135 >=1:8 | 44.8 [31.7 to 58.5] | 18.8 [4.0 to 45.6] | 67.1 [55.6 to 77.3] | 9.5 [1.2 to 30.4]
  Year 5 of study MENACWY-TT-10: hSBA-MenW-135 >=1:8: number analyzed (Participants) | 54 | 14 | 67 | 19
  Year 5 of study MENACWY-TT-10: hSBA-MenW-135 >=1:8 | 44.4 [30.9 to 58.6] | 21.4 [4.7 to 50.8] | 61.2 [48.5 to 72.9] | 26.3 [9.1 to 51.2]
  Year 1 of study MENACWY-TT-10: hSBA-MenY >=1:8: number analyzed (Participants) | 41 | 14 | 89 | 24
  Year 1 of study MENACWY-TT-10: hSBA-MenY >=1:8 | 31.7 [18.1 to 48.1] | 7.1 [0.2 to 33.9] | 65.2 [54.3 to 75.0] | 25.0 [9.8 to 46.7]
  Year 2 of study MENACWY-TT-10: hSBA-MenY >=1:8: number analyzed (Participants) | 56 | 21 | 100 | 27
  Year 2 of study MENACWY-TT-10: hSBA-MenY >=1:8 | 51.8 [38.0 to 65.3] | 33.3 [14.6 to 57.0] | 75.0 [65.3 to 83.1] | 40.7 [22.4 to 61.2]
  Year 3 of study MENACWY-TT-10: hSBA-MenY >=1:8: number analyzed (Participants) | 63 | 21 | 93 | 23
  Year 3 of study MENACWY-TT-10: hSBA-MenY >=1:8 | 50.8 [37.9 to 63.6] | 38.1 [18.1 to 61.6] | 72.0 [61.8 to 80.9] | 34.8 [16.4 to 57.3]
  Year 4 of study MENACWY-TT-10: hSBA-MenY >=1:8: number analyzed (Participants) | 61 | 19 | 84 | 22
  Year 4 of study MENACWY-TT-10: hSBA-MenY >=1:8 | 32.8 [21.3 to 46.0] | 26.3 [9.1 to 51.2] | 67.9 [56.8 to 77.6] | 27.3 [10.7 to 50.2]
  Year 5 of study MENACWY-TT-10: hSBA-MenY >=1:8: number analyzed (Participants) | 58 | 15 | 73 | 18
  Year 5 of study MENACWY-TT-10: hSBA-MenY >=1:8 | 41.4 [28.6 to 55.1] | 40.0 [16.3 to 67.7] | 72.6 [60.9 to 82.4] | 44.4 [21.5 to 69.2]

12. Secondary Outcome: Persistence Phase: Geometric Mean Titers as Measured by hSBA for Each of the 4 Serogroups After 6, 7, 8, 9 and 10 Years of Primary Vaccination
Description: Serogroups included MenA, MenC, MenW-135 and MenY.
Time Frame: 6, 7, 8, 9 and 10 years after primary vaccination (Year 1, 2, 3, 4 and 5 of study MENACWY-TT-100)
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | MenACWY-TT Vaccine: Less Than (<) 2 Years | MenCCRM (Meningitec) Vaccine: Less Than 2 Years | MenACWY-TT Vaccine: Greater Than or Equal to (>=) 2 Years | MenPS (Mencevax ACWY) Vaccine: Less Than 2 Years
Number analyzed (Participants) | 64 | 22 | 100 | 27
titers
  Year 1 of study MENACWY-TT-100: hSBA-MenA: number analyzed (Participants) | 44 | 14 | 90 | 21
  Year 1 of study MENACWY-TT-100: hSBA-MenA | 4.7 [3.2 to 7.1] | 3.5 [2.1 to 5.8] | 6.5 [4.8 to 8.8] | 5.9 [3.0 to 11.7]
  Year 2 of study MENACWY-TT-100: hSBA-MenA: number analyzed (Participants) | 60 | 21 | 99 | 26
  Year 2 of study MENACWY-TT-100: hSBA-MenA | 3.8 [2.9 to 5.2] | 2.8 [1.8 to 4.2] | 4.5 [3.4 to 6.0] | 4.7 [2.4 to 9.0]
  Year 3 of study MENACWY-TT-100: hSBA-MenA: number analyzed (Participants) | 64 | 22 | 97 | 25
  Year 3 of study MENACWY-TT-100: hSBA-MenA | 5.0 [3.5 to 7.1] | 3.7 [2.2 to 6.1] | 4.6 [3.4 to 6.0] | 6.7 [3.2 to 14.0]
  Year 4 of study MENACWY-TT-100: hSBA-MenA: number analyzed (Participants) | 63 | 20 | 86 | 23
  Year 4 of study MENACWY-TT-100: hSBA-MenA | 4.8 [3.5 to 6.6] | 3.4 [2.2 to 5.2] | 6.6 [4.8 to 9.0] | 4.5 [2.4 to 8.8]
  Year 5 of study MENACWY-TT-100: hSBA-MenA: number analyzed (Participants) | 61 | 16 | 69 | 21
  Year 5 of study MENACWY-TT-100: hSBA-MenA | 4.2 [3.1 to 5.9] | 3.1 [2.0 to 4.8] | 4.6 [3.4 to 6.2] | 5.4 [2.5 to 11.7]
  Year 1 of study MENACWY-TT-100: hSBA-MenC: number analyzed (Participants) | 53 | 16 | 97 | 24
  Year 1 of study MENACWY-TT-100: hSBA-MenC | 542.5 [284.8 to 1033.5] | 230.0 [84.3 to 628.1] | 427.2 [260.7 to 700.0] | 234.8 [122.2 to 451.1]
  Year 2 of study MENACWY-TT-100: hSBA-MenC: number analyzed (Participants) | 59 | 20 | 96 | 26
  Year 2 of study MENACWY-TT-100: hSBA-MenC | 368.1 [191.9 to 706.0] | 223.6 [105.8 to 472.7] | 342.7 [200.7 to 585.4] | 169.2 [67.3 to 425.2]
  Year 3 of study MENACWY-TT-100: hSBA-MenC: number analyzed (Participants) | 64 | 22 | 96 | 25
  Year 3 of study MENACWY-TT-100: hSBA-MenC | 378.2 [210.7 to 679.0] | 203.4 [73.8 to 560.9] | 365.5 [214.1 to 624.1] | 273.8 [103.8 to 722.1]
  Year 4 of study MENACWY-TT-100: hSBA-MenC: number analyzed (Participants) | 63 | 20 | 90 | 24
  Year 4 of study MENACWY-TT-100: hSBA-MenC | 319.0 [172.7 to 589.0] | 217.2 [82.8 to 569.9] | 190.4 [112.1 to 323.4] | 125.7 [51.2 to 308.8]
  Year 5 of study MENACWY-TT-100: hSBA-MenC: number analyzed (Participants) | 62 | 16 | 79 | 21
  Year 5 of study MENACWY-TT-100: hSBA-MenC | 362.2 [207.2 to 633.4] | 112.4 [41.2 to 307.0] | 199.3 [118.4 to 335.7] | 119.1 [50.2 to 282.5]
  Year 1 of study MENACWY-TT-100: hSBA-MenW-135: number analyzed (Participants) | 47 | 15 | 92 | 23
  Year 1 of study MENACWY-TT-100: hSBA-MenW-135 | 31.8 [17.5 to 57.8] | 3.3 [1.6 to 6.8] | 62.5 [42.0 to 93.1] | 7.0 [2.9 to 16.9]
  Year 2 of study MENACWY-TT-100: hSBA-MenW-135: number analyzed (Participants) | 58 | 20 | 98 | 27
  Year 2 of study MENACWY-TT-100: hSBA-MenW-135 | 19.5 [11.6 to 32.7] | 4.9 [1.9 to 12.5] | 50.5 [34.5 to 74.1] | 4.0 [2.1 to 7.3]
  Year 3 of study MENACWY-TT-100: hSBA-MenW-135: number analyzed (Participants) | 64 | 21 | 94 | 25
  Year 3 of study MENACWY-TT-100: hSBA-MenW-135 | 8.0 [5.1 to 12.6] | 4.1 [1.9 to 8.6] | 20.4 [13.0 to 32.2] | 3.3 [1.8 to 6.0]
  Year 4 of study MENACWY-TT-100: hSBA-MenW-135: number analyzed (Participants) | 58 | 16 | 79 | 21
  Year 4 of study MENACWY-TT-100: hSBA-MenW-135 | 8.5 [5.3 to 13.5] | 3.7 [1.6 to 8.4] | 23.1 [14.7 to 36.1] | 2.8 [1.7 to 4.4]
  Year 5 of study MENACWY-TT-100: hSBA-MenW-135: number analyzed (Participants) | 54 | 14 | 67 | 19
  Year 5 of study MENACWY-TT-100: hSBA-MenW-135 | 7.6 [4.8 to 11.8] | 3.8 [1.7 to 8.2] | 17.4 [10.8 to 28.0] | 4.2 [2.2 to 8.0]
  Year 1 of study MENACWY-TT-100: hSBA-MenY: number analyzed (Participants) | 41 | 14 | 89 | 24
  Year 1 of study MENACWY-TT-100: hSBA-MenY | 7.9 [4.1 to 15.2] | 3.1 [1.2 to 7.6] | 40.3 [23.9 to 68.1] | 7.3 [2.7 to 19.8]
  Year 2 of study MENACWY-TT-100: hSBA-MenY: number analyzed (Participants) | 56 | 21 | 100 | 27
  Year 2 of study MENACWY-TT-100: hSBA-MenY | 15.8 [9.0 to 27.7] | 6.9 [2.9 to 16.6] | 54.4 [35.0 to 84.4] | 10.5 [4.4 to 25.0]
  Year 3 of study MENACWY-TT-100: hSBA-MenY: number analyzed (Participants) | 63 | 21 | 93 | 23
  Year 3 of study MENACWY-TT-100: hSBA-MenY | 11.6 [7.3 to 18.6] | 8.7 [3.5 to 21.5] | 43.7 [27.5 to 69.5] | 8.8 [3.4 to 22.5]
  Year 4 of study MENACWY-TT-100: hSBA-MenY: number analyzed (Participants) | 61 | 19 | 84 | 22
  Year 4 of study MENACWY-TT-100: hSBA-MenY | 7.3 [4.4 to 11.9] | 5.8 [2.3 to 15.0] | 35.5 [21.5 to 58.8] | 6.2 [2.5 to 15.3]
  Year 5 of study MENACWY-TT-100: hSBA-MenY: number analyzed (Participants) | 58 | 15 | 73 | 18
  Year 5 of study MENACWY-TT-100: hSBA-MenY | 8.6 [5.3 to 14.2] | 8.5 [2.8 to 25.7] | 36.8 [22.4 to 60.7] | 13.9 [4.2 to 46.0]

13. Secondary Outcome: Booster Phase: Percentage of Participants With rSBA Titers >=1:8 and >=1:128 For Each of the 4 Serogroups at 1 Month After Booster Vaccination
Description: Serogroups included MenA, MenC, MenW-135 and MenY.
Time Frame: 1 month after booster vaccination (approximately Year 5.5 of study MENACWY-TT-100)
Population: All eligible participants who received primary vaccination in study MenACWY-TT-027 and booster vaccination in MenACWY-TT-100, had available assay results for 1 month post booster vaccination blood sample. "N": number of participants evaluable for this measure. "Number analyzed": participants analyzed for specified serogroup titers cut off.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MenACWY-TT Vaccine: Less Than (<) 2 Years | MenCCRM (Meningitec) Vaccine: Less Than 2 Years | MenACWY-TT Vaccine: Greater Than or Equal to (>=) 2 Years | MenPS (Mencevax ACWY) Vaccine: Less Than 2 Years
Number analyzed (Participants) | 62 | 16 | 74 | 17
percentage of participants
  rSBA-MenA: >= 1:8 | 98.4 [91.3 to 100.0] | 100.0 [79.4 to 100.0] | 95.9 [88.6 to 99.2] | 100.0 [80.5 to 100.0]
  rSBA-MenC: >= 1:8 | 100.0 [94.2 to 100.0] | 100.0 [79.4 to 100.0] | 100.0 [95.1 to 100.0] | 100.0 [80.5 to 100.0]
  rSBA-MenW-135: >= 1:8: number analyzed (Participants) | 62 | 15 | 74 | 17
  rSBA-MenW-135: >= 1:8 | 100.0 [94.2 to 100.0] | 100.0 [78.2 to 100.0] | 100.0 [95.1 to 100.0] | 94.1 [71.3 to 99.9]
  rSBA-MenY >= 1:8 | 98.4 [91.3 to 100.0] | 100.0 [79.4 to 100.0] | 100.0 [95.1 to 100.0] | 100.0 [80.5 to 100.0]
  rSBA-MenA: >= 1:28 | 98.4 [91.3 to 100.0] | 100.0 [79.4 to 100.0] | 95.9 [88.6 to 99.2] | 100.0 [80.5 to 100.0]
  rSBA-MenC: >= 1:28 | 100.0 [94.2 to 100.0] | 100.0 [79.4 to 100.0] | 100.0 [95.1 to 100.0] | 100.0 [80.5 to 100.0]
  rSBA-MenW-135: >= 1:28: number analyzed (Participants) | 62 | 15 | 74 | 17
  rSBA-MenW-135: >= 1:28 | 100.0 [94.2 to 100.0] | 100.0 [78.2 to 100.0] | 100.0 [95.1 to 100.0] | 94.1 [71.3 to 99.9]
  rSBA-MenY >= 1:28 | 98.4 [91.3 to 100.0] | 100.0 [79.4 to 100.0] | 100.0 [95.1 to 100.0] | 100.0 [80.5 to 100.0]

14. Secondary Outcome: Booster Phase: Geometric Mean Titers as Measured by rSBA For Each of the 4 Serogroups 1 Month After Booster Vaccination
Description: Serogroups included MenA, MenC, MenW-135 and MenY.
Time Frame: 1 month after booster vaccination (approximately Year 5.5 of study MENACWY-TT-100)
Population: All eligible participants who received primary vaccination in study MenACWY-TT-027 and booster vaccination in this study (MenACWY-TT-100) and had available assay results for the 1 month post booster vaccination blood sample. "N": number of participants evaluable for this measure.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | MenACWY-TT Vaccine: Less Than (<) 2 Years | MenCCRM (Meningitec) Vaccine: Less Than 2 Years | MenACWY-TT Vaccine: Greater Than or Equal to (>=) 2 Years | MenPS (Mencevax ACWY) Vaccine: Less Than 2 Years
Number analyzed (Participants) | 62 | 16 | 74 | 17
titers
  rSBA-MenA | 5122.3 [3725.6 to 7042.6] | 4871.0 [2465.1 to 9624.9] | 4626.4 [3040.6 to 7039.4] | 6414.2 [3878.5 to 10607.8]
  rSBA-MenC | 7163.5 [5478.0 to 9367.7] | 5792.6 [3630.6 to 9242.2] | 4020.0 [3319.0 to 4869.1] | 15101.0 [7099.3 to 32121.5]
  rSBA-MenW-135: number analyzed (Participants) | 62 | 15 | 74 | 17
  rSBA-MenW-135 | 25911.2 [19119.7 to 35115.2] | 17970.4 [11666.4 to 27680.7] | 27944.4 [22213.8 to 35153.3] | 10462.5 [3253.5 to 33645.5]
  rSBA-MenY | 7660.5 [5262.9 to 11150.3] | 6316.9 [3223.8 to 12377.5] | 7529.7 [5827.5 to 9729.2] | 6959.2 [3636.7 to 13317.1]

15. Secondary Outcome: Booster Phase: Percentage of Participants With rSBA Booster Response at 1 Month After Booster Vaccination
Description: Serogroups included MenA, MenC, MenW-135 and MenY. rSBA booster response to meningococcal antigens (A,C, W-135 and Y) is defined as: rSBA antibody titer >= 1:32 one month after vaccination, and at least 4-fold increase in rSBA titers one month after vaccination.
Time Frame: 1 month after booster vaccination (approximately Year 5.5 of study MENACWY-TT-100)
Population: All eligible participants who received primary vaccination in study MenACWY-TT-027 and booster vaccination in this study (MenACWY-TT-100), had available assay results for 1 month post booster vaccination blood sample. "N": number of participants evaluable for this measure. "Number analyzed": participants analyzed for specified serogroup.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MenACWY-TT Vaccine: Less Than (<) 2 Years | MenCCRM (Meningitec) Vaccine: Less Than 2 Years | MenACWY-TT Vaccine: Greater Than or Equal to (>=) 2 Years | MenPS (Mencevax ACWY) Vaccine: Less Than 2 Years
Number analyzed (Participants) | 62 | 16 | 74 | 17
percentage of participants
  rSBA-MenA: number analyzed (Participants) | 62 | 16 | 73 | 17
  rSBA-MenA | 90.3 [80.1 to 96.4] | 100.0 [79.4 to 100.0] | 87.7 [77.9 to 94.2] | 94.1 [71.3 to 99.9]
  rSBA-MenC | 82.3 [70.5 to 90.8] | 93.8 [69.8 to 99.8] | 75.7 [64.3 to 84.9] | 94.1 [71.3 to 99.9]
  rSBA-MenW-135: number analyzed (Participants) | 62 | 15 | 74 | 17
  rSBA-MenW-135 | 100.0 [94.2 to 100.0] | 100.0 [78.2 to 100.0] | 100.0 [95.1 to 100.0] | 88.2 [63.6 to 98.5]
  rSBA-MenY | 95.2 [86.5 to 99.0] | 87.5 [61.7 to 98.4] | 93.2 [84.9 to 97.8] | 100.0 [80.5 to 100.0]

16. Secondary Outcome: Booster Phase: Percentage of Participants With hSBA Titers >=1:4 and >=1:8 For Each of the 4 Serogroups at 1 Month After Booster Vaccination
Description: Serogroups included MenA, MenC, MenW-135 and MenY.
Time Frame: 1 month after booster vaccination (approximately Year 5.5 of study MENACWY-TT-100)
Population: All eligible participants: received primary vaccination in study MenACWY-TT-027, booster vaccination in study MenACWY-TT-100, had available assay results for 1 month post booster vaccination blood sample. "N": number of participants evaluable for this measure. "Number analyzed": participants analyzed for specified serogroup titers cut off.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MenACWY-TT Vaccine: Less Than (<) 2 Years | MenCCRM (Meningitec) Vaccine: Less Than 2 Years | MenACWY-TT Vaccine: Greater Than or Equal to (>=) 2 Years | MenPS (Mencevax ACWY) Vaccine: Less Than 2 Years
Number analyzed (Participants) | 62 | 16 | 74 | 17
percentage of participants
  hSBA-MenA: >=1:4: number analyzed (Participants) | 62 | 16 | 73 | 17
  hSBA-MenA: >=1:4 | 100.0 [94.2 to 100.0] | 87.5 [61.7 to 98.4] | 100.0 [95.1 to 100.0] | 100.0 [80.5 to 100.0]
  hSBA-MenC: >=1:4: number analyzed (Participants) | 59 | 15 | 71 | 17
  hSBA-MenC: >=1:4 | 100.0 [93.9 to 100.0] | 100.0 [78.2 to 100.0] | 100.0 [94.9 to 100.0] | 94.1 [71.3 to 99.9]
  hSBA-MenW-135: >=1:4: number analyzed (Participants) | 62 | 13 | 74 | 15
  hSBA-MenW-135: >=1:4 | 100.0 [94.2 to 100.0] | 100.0 [75.3 to 100.0] | 100.0 [95.1 to 100.0] | 100.0 [78.2 to 100.0]
  hSBA-MenY: >=1:4: number analyzed (Participants) | 61 | 15 | 74 | 17
  hSBA-MenY: >=1:4 | 100.0 [94.1 to 100.0] | 93.3 [68.1 to 99.8] | 100.0 [95.1 to 100.0] | 100.0 [80.5 to 100.0]
  hSBA-MenA: >=1:8: number analyzed (Participants) | 62 | 16 | 73 | 17
  hSBA-MenA: >=1:8 | 100.0 [94.2 to 100.0] | 87.5 [61.7 to 98.4] | 100.0 [95.1 to 100.0] | 100.0 [80.5 to 100.0]
  hSBA-MenC: >=1:8: number analyzed (Participants) | 59 | 15 | 71 | 17
  hSBA-MenC: >=1:8 | 100.0 [93.9 to 100.0] | 100.0 [78.2 to 100.0] | 100.0 [94.9 to 100.0] | 94.1 [71.3 to 99.9]
  hSBA-MenW-135: >=1:8: number analyzed (Participants) | 62 | 13 | 74 | 15
  hSBA-MenW-135: >=1:8 | 100.0 [94.2 to 100.0] | 100.0 [75.3 to 100.0] | 100.0 [95.1 to 100.0] | 100.0 [78.2 to 100.0]
  hSBA-MenY: >=1:8: number analyzed (Participants) | 61 | 15 | 74 | 17
  hSBA-MenY: >=1:8 | 100.0 [94.1 to 100.0] | 93.3 [68.1 to 99.8] | 100.0 [95.1 to 100.0] | 100.0 [80.5 to 100.0]

17. Secondary Outcome: Booster Phase: Geometric Mean Titers Using hSBA For Each of the 4 Serogroups at 1 Month After Booster Vaccination
Description: Serogroups included MenA, MenC, MenW-135 and MenY.
Time Frame: 1 month after booster vaccination (approximately Year 5.5 of study MENACWY-TT-100)
Population: as for outcome 16
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | MenACWY-TT Vaccine: Less Than (<) 2 Years | MenCCRM (Meningitec) Vaccine: Less Than 2 Years | MenACWY-TT Vaccine: Greater Than or Equal to (>=) 2 Years | MenPS (Mencevax ACWY) Vaccine: Less Than 2 Years
Number analyzed (Participants) | 62 | 16 | 74 | 17
titers
  hSBA-MenA: number analyzed (Participants) | 62 | 16 | 73 | 17
  hSBA-MenA | 1534.2 [1112.1 to 2116.6] | 90.0 [35.7 to 227.1] | 1213.0 [993.9 to 1480.5] | 211.1 [130.9 to 340.3]
  hSBA-MenC: number analyzed (Participants) | 59 | 15 | 71 | 17
  hSBA-MenC | 33959.8 [23890.2 to 48273.5] | 42559.2 [20106.2 to 90086.2] | 15543.5 [11734.9 to 20588.3] | 44794.4 [10111.6 to 198440.4]
  hSBA-MenW-135: number analyzed (Participants) | 62 | 13 | 74 | 15
  hSBA-MenW-135 | 11924.8 [8715.6 to 16315.7] | 258.1 [155.7 to 427.8] | 6965.2 [5274.3 to 9198.3] | 199.6 [101.0 to 394.7]
  hSBA-MenY: number analyzed (Participants) | 61 | 15 | 74 | 17
  hSBA-MenY | 12154.3 [9660.9 to 15291.1] | 407.8 [129.9 to 1280.3] | 11127.4 [8909.2 to 13898.0] | 453.9 [214.6 to 959.8]

18. Secondary Outcome: Booster Phase: Percentage of Participants With hSBA Booster Response at 1 Month After Booster Vaccination
Description: Serogroups included MenA, MenC, MenW-135 and MenY. hSBA booster response to meningococcal antigens (A,C, W-135 and Y) is defined as: hSBA antibody titer >= 1:8 one month after vaccination, and at least 4-fold increase in hSBA titers one month after vaccination.
Time Frame: 1 month after booster vaccination (approximately Year 5.5 of study MENACWY-TT-100)
Population: All eligible participants: received primary vaccination in study MenACWY-TT-027, booster vaccination in study MenACWY-TT-100, had available assay results for 1 month post booster vaccination blood sample. "N": number of participants evaluable for this measure. "Number analyzed": participants analyzed for specified serogroup.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MenACWY-TT Vaccine: Less Than (<) 2 Years | MenCCRM (Meningitec) Vaccine: Less Than 2 Years | MenACWY-TT Vaccine: Greater Than or Equal to (>=) 2 Years | MenPS (Mencevax ACWY) Vaccine: Less Than 2 Years
Number analyzed (Participants) | 59 | 15 | 70 | 17
percentage of participants
  hSBA-MenA: number analyzed (Participants) | 59 | 15 | 61 | 17
  hSBA-MenA | 98.3 [90.9 to 100.0] | 93.3 [68.1 to 99.8] | 100.0 [94.1 to 100.0] | 88.2 [63.6 to 98.5]
  hSBA-MenC: number analyzed (Participants) | 57 | 14 | 70 | 17
  hSBA-MenC | 86.0 [74.2 to 93.7] | 92.9 [66.1 to 99.8] | 85.7 [75.3 to 92.9] | 94.1 [71.3 to 99.9]
  hSBA-MenW-135: number analyzed (Participants) | 52 | 11 | 59 | 14
  hSBA-MenW-135 | 100.0 [93.2 to 100.0] | 90.9 [58.7 to 99.8] | 96.6 [88.3 to 99.6] | 100.0 [76.8 to 100.0]
  hSBA-MenY: number analyzed (Participants) | 56 | 14 | 65 | 14
  hSBA-MenY | 100.0 [93.6 to 100.0] | 71.4 [41.9 to 91.6] | 98.5 [91.7 to 100.0] | 78.6 [49.2 to 95.3]

19. Secondary Outcome: Persistence Phase: Percentage of Participants With Serious Adverse Events (SAEs) Related to Vaccination or Any Adverse Event (AE) Related to Lack of Vaccine Efficacy
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs related to "lack of vaccine efficacy" were as judged by the investigator.
Time Frame: Through 5 years (6, 7, 8, 9 and 10 years post primary vaccination)
Population: All the participants enrolled in the study.
Measure: Number; unit: percentage of participants
Arm/Group | MenACWY-TT Vaccine: Less Than (<) 2 Years | MenCCRM (Meningitec) Vaccine: Less Than 2 Years | MenACWY-TT Vaccine: Greater Than or Equal to (>=) 2 Years | MenPS (Mencevax ACWY) Vaccine: Less Than 2 Years
Number analyzed (Participants) | 76 | 23 | 115 | 29
percentage of participants | 0.0 | 0.0 | 0.0 | 0.0

20. Secondary Outcome: Booster Phase: Percentage of Participants With Solicited Local and General Adverse Events up to 4 Days Post Booster Vaccination
Description: Solicited general events: fatigue, gastrointestinal (GI) events (nausea, vomiting, diarrhea and/or abdominal pain, headache (0= normal, 1=mild/easily tolerated, 2=moderate/interfered with normal activity, 3=severe/prevented normal activity) and fever (>=37.5°C for oral/axillary/tympanic route, >=38.0°C for rectal route). Solicited local events: pain (0=none, 1=mild, not interfered/prevented normal activity, 2=moderate, painful when limb moved/interfered with normal activity, 3=severe, significant pain at rest/prevented normal activity), redness and swelling at injection site (record greatest surface diameter in millimeter (mm) as 0 to <=20 mm, >20 to <=50 mm, >50 mm). Participants may be represented in more than 1 category. Only categories with at least 1 participant reported. 'Medical advice' signifies medical advice received to resolve any event. 'Related'=relationship to study vaccine assessed by investigator.
Time Frame: Up to 4 days post booster vaccination
Population: Analysis population included all participants who received a booster dose of study vaccine MenACWY-TT in the booster stage. "Number analyzed": participants analyzed for specified category.
Measure: Number; unit: percentage of participants
Arm/Group | MenACWY-TT Vaccine: Less Than (<) 2 Years | MenCCRM (Meningitec) Vaccine: Less Than 2 Years | MenACWY-TT Vaccine: Greater Than or Equal to (>=) 2 Years | MenPS (Mencevax ACWY) Vaccine: Less Than 2 Years
Number analyzed (Participants) | 67 | 16 | 77 | 21
percentage of participants
  All pain: number analyzed (Participants) | 67 | 16 | 74 | 21
  All pain | 59.7 | 56.3 | 59.5 | 61.9
  Pain: Grade 1: number analyzed (Participants) | 67 | 16 | 74 | 21
  Pain: Grade 1 | 43.3 | 37.5 | 40.5 | 42.9
  Pain: Grade 2: number analyzed (Participants) | 67 | 16 | 74 | 21
  Pain: Grade 2 | 16.4 | 18.8 | 16.2 | 19.0
  Severe pain: Grade 3: number analyzed (Participants) | 67 | 16 | 74 | 21
  Severe pain: Grade 3 | 0.0 | 0.0 | 2.7 | 0.0
  All redness: number analyzed (Participants) | 67 | 16 | 74 | 21
  All redness | 35.8 | 43.8 | 36.5 | 23.8
  Redness: 0 to <=20 mm: number analyzed (Participants) | 67 | 16 | 74 | 21
  Redness: 0 to <=20 mm | 28.4 | 25.0 | 31.1 | 14.3
  Redness: >20 to <=50 mm: number analyzed (Participants) | 67 | 16 | 74 | 21
  Redness: >20 to <=50 mm | 1.5 | 18.8 | 2.7 | 0.0
  Redness: >50 mm: number analyzed (Participants) | 67 | 16 | 74 | 21
  Redness: >50 mm | 6.0 | 0.0 | 2.7 | 9.5
  All swelling | 17.9 | 6.3 | 23.0 | 14.3
  Swelling: 0 to <=20 mm: number analyzed (Participants) | 67 | 16 | 74 | 21
  Swelling: 0 to <=20 mm | 14.9 | 0.0 | 16.2 | 0.0
  Swelling: >20 to <=50 mm: number analyzed (Participants) | 67 | 16 | 74 | 21
  Swelling: >20 to <=50 mm | 1.5 | 6.3 | 1.4 | 4.8
  Swelling: >50 mm: number analyzed (Participants) | 67 | 16 | 74 | 21
  Swelling: >50 mm | 1.5 | 0.0 | 5.4 | 9.5
  All fatigue: number analyzed (Participants) | 67 | 16 | 74 | 21
  All fatigue | 31.3 | 12.5 | 29.7 | 23.8
  Fatigue: Grade 1: number analyzed (Participants) | 67 | 16 | 74 | 21
  Fatigue: Grade 1 | 20.9 | 12.5 | 16.2 | 14.3
  Fatigue: Grade 2: number analyzed (Participants) | 67 | 16 | 74 | 21
  Fatigue: Grade 2 | 9.0 | 0.0 | 6.8 | 9.5
  Fatigue: Grade 3: number analyzed (Participants) | 67 | 16 | 74 | 21
  Fatigue: Grade 3 | 1.5 | 0.0 | 6.8 | 0.0
  Fatigue: Related fatigue: number analyzed (Participants) | 67 | 16 | 74 | 21
  Fatigue: Related fatigue | 31.3 | 12.5 | 29.7 | 23.8
  Fatigue: Grade 3 Related: number analyzed (Participants) | 67 | 16 | 74 | 21
  Fatigue: Grade 3 Related | 1.5 | 0.0 | 6.8 | 0.0
  All fever: number analyzed (Participants) | 67 | 16 | 74 | 21
  All fever | 1.5 | 0.0 | 0.0 | 0.0
  Fever: Grade 1: number analyzed (Participants) | 67 | 16 | 74 | 21
  Fever: Grade 1 | 1.5 | 0.0 | 0.0 | 0.0
  Fever: Grade 2: number analyzed (Participants) | 67 | 16 | 74 | 21
  Fever: Grade 2 | 0.0 | 0.0 | 0.0 | 0.0
  Fever: Grade 3: number analyzed (Participants) | 67 | 16 | 74 | 21
  Fever: Grade 3 | 0.0 | 0.0 | 0.0 | 0.0
  Fever: Related: number analyzed (Participants) | 67 | 16 | 74 | 21
  Fever: Related | 1.5 | 0.0 | 0.0 | 0.0
  Fever: Grade 3 related: number analyzed (Participants) | 67 | 16 | 74 | 21
  Fever: Grade 3 related | 0.0 | 0.0 | 0.0 | 0.0
  All gastrointestinal event (GI): number analyzed (Participants) | 67 | 16 | 74 | 21
  All gastrointestinal event (GI) | 9.0 | 0.0 | 17.6 | 14.3
  GI: Grade 1: number analyzed (Participants) | 67 | 16 | 74 | 21
  GI: Grade 1 | 7.5 | 0.0 | 13.5 | 4.8
  GI: Grade 2: number analyzed (Participants) | 67 | 16 | 74 | 21
  GI: Grade 2 | 1.5 | 0.0 | 2.7 | 9.5
  GI: Grade 3: number analyzed (Participants) | 67 | 16 | 74 | 21
  GI: Grade 3 | 0.0 | 0.0 | 1.4 | 0.0
  GI: Related: number analyzed (Participants) | 67 | 16 | 74 | 21
  GI: Related | 7.5 | 0.0 | 17.6 | 14.3
  GI: Grade 3 related: number analyzed (Participants) | 67 | 16 | 74 | 21
  GI: Grade 3 related | 0.0 | 0.0 | 1.4 | 0.0
  All headache: number analyzed (Participants) | 67 | 16 | 74 | 21
  All headache | 20.9 | 31.3 | 27.0 | 23.8
  Headache: Grade 1: number analyzed (Participants) | 67 | 16 | 74 | 21
  Headache: Grade 1 | 14.9 | 18.8 | 18.9 | 19.0
  Headache: Grade 2: number analyzed (Participants) | 67 | 16 | 74 | 21
  Headache: Grade 2 | 6.0 | 12.5 | 6.8 | 4.8
  Headache: Grade 3: number analyzed (Participants) | 67 | 16 | 74 | 21
  Headache: Grade 3 | 0.0 | 0.0 | 1.4 | 0.0
  Headache: Related: number analyzed (Participants) | 67 | 16 | 74 | 21
  Headache: Related | 17.9 | 31.3 | 24.3 | 23.8
  Headache: Grade 3 related: number analyzed (Participants) | 67 | 16 | 74 | 21
  Headache: Grade 3 related | 0.0 | 0.0 | 1.4 | 0.0
  Headache: Medical advice: number analyzed (Participants) | 67 | 16 | 74 | 21
  Headache: Medical advice | 0.0 | 0.0 | 1.4 | 0.0

21. Secondary Outcome: Booster Phase: Percentage of Participants With Unsolicited Adverse Events up to 31 Days Post Booster Vaccination
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An unsolicited AE covers any untoward medical occurrence in a clinical investigation participant temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Time Frame: Up to 31 days post booster vaccination
Population: Analysis population included all participants who received a booster dose of study vaccine MenACWY-TT in the booster stage.
Measure: Number; unit: percentage of participants
Arm/Group | MenACWY-TT Vaccine: Less Than (<) 2 Years | MenCCRM (Meningitec) Vaccine: Less Than 2 Years | MenACWY-TT Vaccine: Greater Than or Equal to (>=) 2 Years | MenPS (Mencevax ACWY) Vaccine: Less Than 2 Years
Number analyzed (Participants) | 67 | 16 | 77 | 21
percentage of participants | 23.9 | 31.3 | 35.1 | 52.4

22. Secondary Outcome: Booster Phase: Percentage of Participants With Serious Adverse Events (SAEs) Up to 6 Months Post Booster Vaccination
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Up to 6 months post booster vaccination
Population: as for outcome 21
Measure: Number; unit: percentage of participants
Arm/Group | MenACWY-TT Vaccine: Less Than (<) 2 Years | MenCCRM (Meningitec) Vaccine: Less Than 2 Years | MenACWY-TT Vaccine: Greater Than or Equal to (>=) 2 Years | MenPS (Mencevax ACWY) Vaccine: Less Than 2 Years
Number analyzed (Participants) | 67 | 16 | 77 | 21
percentage of participants | 0.0 | 0.0 | 1.3 | 0.0

23. Secondary Outcome: Booster Phase: Percentage of Participants With New Onset Chronic Illness Up to 6 Months Post Booster Vaccination
Description: New onset chronic illness included autoimmune disorders, asthma, type I diabetes, allergies.
Time Frame: Up to 6 months post booster vaccination
Population: as for outcome 21
Measure: Number; unit: percentage of participants
Arm/Group | MenACWY-TT Vaccine: Less Than (<) 2 Years | MenCCRM (Meningitec) Vaccine: Less Than 2 Years | MenACWY-TT Vaccine: Greater Than or Equal to (>=) 2 Years | MenPS (Mencevax ACWY) Vaccine: Less Than 2 Years
Number analyzed (Participants) | 67 | 16 | 77 | 21
percentage of participants | 0.0 | 0.0 | 1.3 | 4.8

ADVERSE EVENTS:
Time Frame: For persistence phase: Through 5 years (6, 7, 8, 9 and 10 years post primary vaccination); Booster phase: up to 6 months after booster vaccination
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event.
Groups:
- Persistence Phase: MenACWY-TT Vaccine (Less Than [<] 2 Years): Participants with <2 years of age, received a single 0.5 mL dose of MenACWY-TT vaccine intramuscularly, as primary vaccination in study MENACWY-TT-027. Then, in this study they were evaluated for long-term persistence for a maximum duration of 5 years (6, 7, 8, 9 and 10 years post primary vaccination in MENACWY-TT-027).
- Persistence Phase:MenCCRM (Meningitec) Vaccine(<2 Years): Participants with <2 years of age, received a single 0.5 mL dose of Meningitec vaccine intramuscularly, as primary vaccination in study MENACWY-TT-027. Then, in this study they were evaluated for long-term persistence for a maximum duration of 5 years (6, 7, 8, 9 and 10 years post primary vaccination in MENACWY-TT-027).
- Persistence Phase: MenACWY-TT Vaccine (>=2 Years): Participants with >=2 years of age, received a single 0.5 mL dose of MenACWY-TT vaccine intramuscularly, as primary vaccination in study MENACWY-TT-027. Then, in this study they were evaluated for long-term persistence for a maximum duration of 5 years (6, 7, 8, 9 and 10 years post primary vaccination in MENACWY-TT-027).
- Persistence Phase: MenPS (Mencevax ACWY) Vaccine (< 2 Years): Participants with <2 years of age, received a single 0.5 mL dose of MencevaxACWY vaccine intramuscularly, as primary vaccination in study MENACWY-TT-027. Then, in this study they were evaluated for long term persistence for a maximum duration of 5 years (6, 7, 8, 9 and 10 years post primary vaccination in MENACWY-TT-027).
- Booster Phase: MenACWY-TT Vaccine (Less Than 2 Years): Persistence phase: Participants with <2 years of age, received a single 0.5 mL dose of MenACWY-TT vaccine intramuscularly, as primary vaccination in study MENACWY-TT-027. Then, in this study they were evaluated for long-term persistence for a maximum duration of 5 years (6, 7, 8, 9 and 10 years post primary vaccination in MENACWY-TT-027). Booster phase: Participants received a single 0.5 mL booster dose of MenACWY-TT intramuscularly in this study, 10 years post primary vaccination in MENACWY-TT-027, and were followed up for 6 months.
- Booster Phase: MenCCRM (Meningitec) Vaccine (<2 Years): Persistence phase: Participants with <2 years of age, received a single 0.5 mL dose of Meningitec vaccine intramuscularly, as primary vaccination in study MENACWY-TT-027. Then, in this study they were evaluated for long-term persistence for a maximum duration of 5 years (6, 7, 8, 9 and 10 years post primary vaccination in MENACWY-TT-027). Booster phase: Participants received a single 0.5 mL booster dose of MenACWY-TT intramuscularly in this study, 10 years post primary vaccination, and were followed up for 6 months.
- Booster Phase: MenACWY-TT Vaccine (>= 2 Years): Persistence phase: Participants with >=2 years of age, received a single 0.5 mL dose of MenACWY-TT vaccine intramuscularly, as primary vaccination in study MENACWY-TT-027. Then, in this study they were evaluated for long-term persistence for a maximum duration of 5 years (6, 7, 8, 9 and 10 years post primary vaccination in MENACWY-TT-027). Booster phase: Participants received a single 0.5 mL booster dose of MenACWY-TT in this study, 10 years post primary vaccination, and were followed up for 6 months.
- Booster Phase: MenPS (Mencevax ACWY) Vaccine (<2 Years): Persistence phase: Participants with <2 years of age, received a single 0.5 mL dose of MencevaxACWY vaccine intramuscularly, as primary vaccination in study MENACWY-TT-027. Then, in this study they were evaluated for long term persistence for a maximum duration of 5 years (6, 7, 8, 9 and 10 years post primary vaccination in MENACWY-TT-027). Booster phase: Participants received a single 0.5 mL booster dose of MenACWY-TT in this study, 10 years post primary vaccination, and were followed up for 6 months.
Arm/Group | Persistence Phase: MenACWY-TT Vaccine (Less Than [<] 2 Years) | Persistence Phase:MenCCRM (Meningitec) Vaccine(<2 Years) | Persistence Phase: MenACWY-TT Vaccine (>=2 Years) | Persistence Phase: MenPS (Mencevax ACWY) Vaccine (< 2 Years) | Booster Phase: MenACWY-TT Vaccine (Less Than 2 Years) | Booster Phase: MenCCRM (Meningitec) Vaccine (<2 Years) | Booster Phase: MenACWY-TT Vaccine (>= 2 Years) | Booster Phase: MenPS (Mencevax ACWY) Vaccine (<2 Years)
All-Cause Mortality (participants affected / at risk) | 0/76 | 0/23 | 0/115 | 0/29 | 0/67 | 0/16 | 0/77 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/76 | 0/23 | 0/115 | 0/29 | 0/67 | 0/16 | 1/77 | 0/21
Other Adverse Events (participants affected / at risk) | 0/76 | 0/23 | 0/115 | 0/29 | 53/67 | 12/16 | 65/77 | 15/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Persistence Phase: MenACWY-TT Vaccine (Less Than [<] 2 Years) (N=76) | Persistence Phase:MenCCRM (Meningitec) Vaccine(<2 Years) (N=23) | Persistence Phase: MenACWY-TT Vaccine (>=2 Years) (N=115) | Persistence Phase: MenPS (Mencevax ACWY) Vaccine (< 2 Years) (N=29) | Booster Phase: MenACWY-TT Vaccine (Less Than 2 Years) (N=67) | Booster Phase: MenCCRM (Meningitec) Vaccine (<2 Years) (N=16) | Booster Phase: MenACWY-TT Vaccine (>= 2 Years) (N=77) | Booster Phase: MenPS (Mencevax ACWY) Vaccine (<2 Years) (N=21)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Persistence Phase: MenACWY-TT Vaccine (Less Than [<] 2 Years) (N=76) | Persistence Phase:MenCCRM (Meningitec) Vaccine(<2 Years) (N=23) | Persistence Phase: MenACWY-TT Vaccine (>=2 Years) (N=115) | Persistence Phase: MenPS (Mencevax ACWY) Vaccine (< 2 Years) (N=29) | Booster Phase: MenACWY-TT Vaccine (Less Than 2 Years) (N=67) | Booster Phase: MenCCRM (Meningitec) Vaccine (<2 Years) (N=16) | Booster Phase: MenACWY-TT Vaccine (>= 2 Years) (N=77) | Booster Phase: MenPS (Mencevax ACWY) Vaccine (<2 Years) (N=21)
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Coeliac disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal symptoms (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 6 | 0 | 13 | 3
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Axillary pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Fatigue 1 (General disorders) | 0 | 0 | 0 | 0 | 21 | 2 | 22 | 5
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Injection site bruising (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Injection site erythema (redness) (General disorders) | 0 | 0 | 0 | 0 | 24 | 7 | 27 | 5
Injection site hypoaesthesia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection site pain (pain at injection site) (General disorders) | 0 | 0 | 0 | 0 | 40 | 9 | 44 | 13
Injection site pruritus (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Injection site swelling (swelling) (General disorders) | 0 | 0 | 0 | 0 | 12 | 1 | 17 | 3
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Hand-foot-and-mouth disease (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infectious mononucleosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 7 | 2
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache 1 (Nervous system disorders) | 0 | 0 | 0 | 0 | 14 | 5 | 20 | 5
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 4 | 1 | 3 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2016-02-25): https://cdn.clinicaltrials.gov/large-docs/07/NCT01962207/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-26): https://cdn.clinicaltrials.gov/large-docs/07/NCT01962207/SAP_001.pdf